CLINICAL TRIAL: NCT01559142
Title: Efficacy and Safety of Induction Therapy With Three Doses of Infliximab in Patients With Crohn Disease Aged 7-17 Years-multicenter Open Study. Efficacy and Safety of Two Regimens of Maintenance Therapy in Patients With Crohn Disease Aged 7-17 Years-multicenter Randomized Study
Brief Title: Efficacy and Safety of Two Regimens of Maintenance Therapy in Children With Crohn Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Memorial Health Institute, Poland (Other)
Responsible Party: Principal Investigator, JAROSLAW KIERKUS, MD, PhD, Children's Memorial Health Institute, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP CZD 2008-01-14
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; infliximab; azathioprine
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IFX TG (Active Comparator)
  Interventions: Drug: Infliximab with azathioprine (IIFX + AZA)
- IFX alone (Active Comparator)
  Interventions: Drug: Infliximab (IFX alone)

INTERVENTIONS:
Drug: Infliximab with azathioprine (IIFX + AZA) — Infliximab with azathioprine during whole one year study
  Arms: IFX TG
Drug: Infliximab (IFX alone) — Infliximab continuously; azathioprine stopped in 26 week
  Arms: IFX alone

SUMMARY:
The aim of the study is confirmation of efficacy of induction therapy with three doses of infliximab In patients with Crohn disease aged 7-17 years, and comparison of efficacy and safety of two regiment of maintenance therapy:

1. Infliximab with immunomodulation
2. Infliximab alone

DETAILED DESCRIPTION:
Study project Screening (Days -14 do 0): Laboratory and endoscopic (up to three months before Day 0) results will be obtained to check with inclusion/exclusion criteria.

Part A (Days 1 to 71): Induction therapy with 3 doses of infliximab 5 mg/kg will be applied on days 1 - 15 - 43. Simultaneously in patients receiving steroids, steroid tapering will be performed up to 71 Day. At Day 71 clinical (PCDAI) and endoscopic assessment will be done. Patients with no clinical response will be qualified to Follow-up surveillance group. Patients with clinical response present will be randomized to two groups of maintenance therapy:

1. Infliximab with immunomodulation 2. Infliximab alone

Part B (Weeks 10 - 54): Patient with both groups will have scheduled visits at Weeks 14, 22, 30, 38, 46. Infliximab infusions and laboratory tests will be performed at each visit. At Week 54 clinical (PCDAI) and endoscopic assessment will be done.

Follow Up: 4 weeks after last visit - SAE monitoring Aim of the study

The aim of the study is confirmation of efficacy of induction therapy with three doses of infliximab In patients with Crohn disease aged 7-17 years, and comparison of efficacy and safety of two regiment of maintenance therapy:

1. Infliximab with immunomodulation
2. Infliximab alone Drug dosing in therapy regimens.

   Infliximab: 5 mg/kg mc In intravenous infusion lasting over 2 hrs. Azathioprine: 1,5 - 3 mg/kg/24h Methotrexate: 10 - 25 mg/week

   Safety assessment

   AE and SAE monitoring will be conducted during whole period of the study

   Efficacy assessment

   Primary endpoint

   Part A:

   • Clinical response defined as: Decrease of PCDAI ≥ 15 points AND PCDAI less than 30 points

   • Remission defined as: PCDAI ≤ 10 points

   Part B:
   * Loss of clinical response defined as:

   Increase of PCDAI more than 15 points OR PCDAI > 30 points

   Secondary endpoints

   Part A:

   • Time to steroid cessation

   Part B:

   • Necessity to increase/change maintenance therapy with

   o Surgery

   o Increase of infliximab dose
   * Increase of immunomodulator dose
   * Steroids induction

   Statistical methods
   * ITT analysis
   * Primary endpoints: chi2 tests, Kaplan-Meier analysis
   * Secondary endpoints: chi2 tests, Kaplan-Meier analysis, U Mann-Whitney analysis

ELIGIBILITY:
Inclusion Criteria:

1. Patients with severe Crohn disease (PCDAI in anamnesis more than 51 points), with PCDAI currently over 30 points, with no or loss of response for previous therapy (except biological agents). Patients may have active fistulas.
2. Efficient methods of contraception in patients of childbearing potential during study period and six months after.
3. Patients will be enrolled to Part B of the study whether they finish Part A with clinical remission or clinical response.

Exclusion Criteria:

1. Hypersensitivity to infliximab
2. Pregnancy and breastfeeding
3. Active tuberculosis or other severe infection: sepsis, opportunistic infections, active CMV, yersinia pseudotuberculosis, pneumocystis carini, atypical mycobacteriosis
4. VZV infection, hepatitis, pneumonia during 3 months before Day 0 of the study
5. pancytopaenia and aplastic anemia
6. moderate and severe heart insufficiency (NYHA class III/IV), or unstable coronary heart disease
7. chronic pulmonary insufficiency, chronic renal insufficiency, chronic liver insufficiency
8. HIV infection
9. Presence of severe diseases of nervous system or severe endocrinological, hematological, psychiatric diseases.
10. Demyelinisation syndrome or symptoms resembling Demyelinisation syndrome
11. Malignancy or premalignant conditions during 5 years before Day 0 of the study.
12. Severe infection currently present
13. Malignancy currently present

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2008-11; Primary Completion 2012-04 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Clinical disease activity | 14 week and one year

SECONDARY OUTCOMES:
endoscopic disease activity | 14 week and one year

CONTACTS AND LOCATIONS:
Overall Officials: Jaroslaw Kierkus, MD PhD, Principal Investigator — The Children's Memorial Institute
Locations (1):
- Department of Gastroenterology, Hepatology and Feeding Disorders, Warsaw, Poland